CLINICAL TRIAL: NCT00615641
Title: Relationship of Dietary Factors and Physical Activity to Body Fat in 3-5 Year Old Children
Brief Title: Diet, Exercise and Body Fat in 3-5 Year Olds
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: University of Arkansas (Other); United States Department of Agriculture (USDA) (U.S. Federal Agency); Life Measurement Inc. (Industry); Texas Woman's University (Other)
Responsible Party: Tina Crook, M.S., R.D. / Principal Investigator, Arkansas Children's Nutrition Center
Other Study IDs: 72850; CRIS # 6251-51000-005-03S
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-02

CONDITIONS: Healthy
Keywords: Children; Nutrition; Body Fat; Physical Activity; Diet; Childhood Obesity; Healthy Children
MeSH Terms: conditions — Motor Activity; Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: 3 year old children
- 2: 4 year old children
- 3: 5 year old children

SUMMARY:
To determine how practical and precise different body composition methods are for measuring body fat and lean tissue in young children and to determine if certain dietary factors and physical activity patterns are related to body fat in children.

ELIGIBILITY:
Inclusion Criteria:

* 3-5 year old children
* Full term at birth
* English as primary language
* Weighed at least 5.5# at birth
* Parent or guardian is at least 18 years of age

Exclusion Criteria:

* Child has any chronic condition, metabolic disorder, pulmonary disorder, bone disorder, condition that may affect growth, ADD or ADHD
* Child on any medication thought to interfere with study parameters as determined by the investigator

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: We are seeking healthy 3-5 year old children in the greater Little Rock area.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2007-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tina Crook, M.S., R.D., Principal Investigator — Arkansas Children's Nutrition Center
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States